CLINICAL TRIAL: NCT00914940
Title: A Multi-center Phase II Study of Selective Depletion of CD45RA+ T Cells From Allogeneic Peripheral Blood Stem Cell Grafts for the Prevention of GVHD
Brief Title: Selective Depletion of CD45RA+T Cells From Allogeneic Peripheral Blood Stem Cell Grafts for the Prevention of GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not reach one of the primary endpoints of decreased total acute GVHD
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2222.00; P30CA015704 (NIH); P01CA018029 (NIH); IR-6907 (Other: FHCRC IRB); CDR0000644201 (Registry Identifier: NCI PDQ); 0903004832 (Other: HIC Protocol Number); NCI-2010-00713 (Registry Identifier: NCI / CTRP); RG2810004 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-07

CONDITIONS: Graft Versus Host Disease; Leukemia; Myelodysplastic Syndromes
Keywords: graft versus host disease; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; childhood acute lymphoblastic leukemia in remission; recurrent childhood acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute myeloid leukemia in remission; recurrent childhood acute myeloid leukemia; childhood myelodysplastic syndromes; previously treated myelodysplastic syndromes; refractory anemia with excess blasts; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Congenital Abnormalities; Anemia, Refractory, with Excess of Blasts | interventions — fludarabine phosphate; Tacrolimus; Thiotepa; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): CONDITIONING: Patients undergo total-body irradiation twice daily on days -10 to -7. Patients also receive thiotepa IV over 4 hours on days -6 and -5 and fludarabine IV over 30 minutes on days -6 to -2. TRANSPLANTATION: Patients undergo infusion of CD34+ enriched allogeneic peripheral blood stem cells (PBSC) followed by CD45RA+ T-cell-depleted allogeneic PBSC on day 0.
  GRAFT-VS-HOST DISEASE PROPHYLAXIS: Cohort A: Patients receive tacrolimus IV continuously or orally twice daily beginning on day -1 and continuing until day 50 followed by standard taper in the absence of grade II-IV acute GVHD. Cohort B: Patients receive tacrolimus IV continuously or orally twice daily beginning on day -1 and continuing until day 30 followed by rapid taper in the absence of grade II-IV acute GVHD.
  Interventions: Drug: Fludarabine Phosphate; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation (TBI); Other: Magnetic Affinity Cell Sorting; Procedure: Peripheral Blood Stem Cell Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: Fludarabine Phosphate — Fludarabine will be administered in a dose of 25 mg/m2/day IV over approximately 30 minutes for 5 consecutive days (day -6 to -2). The total dose of fludarabine will be 125 mg/m2.
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: Tacrolimus — Tacrolimus will be administered beginning on day -1 at a dose of 0.03 mg/kg/day by continuous IV infusion.
  For the first cohort of 35 patients, if there is no evidence of grade II-IV acute GVHD on or prior to day 50, tacrolimus should then be tapered at the rate of approximately 5% of the day 50 dose each week for liquid, and 20% of the day 50 dose per month for capsules.
  In the second cohort of 25 patients if there is no evidence of grade II GVHD on or prior to day 30, tacrolimus should then be tapered at the rate of approximately 8% of the day 30 dose each week for liquid, and 33% of the day 30 dose per month for capsules.
  Other Names: Advagraf; FK 506; Prograf; Protopic
Drug: Thiotepa — Thiotepa will be administered in a dose of 5 mg/kg/day (adjusted body weight) IV over approximately 4 hours for 2 consecutive days (day -6 and day -5).
  Other Names: Oncotiotepa; STEPA; TESPA; Tespamin; Tespamine; TSPA
Radiation: Total-Body Irradiation (TBI) — TBI will be given as 165 cGy fractions twice per day x 4 days - total dose 1320cGy (days -10 to -7).
  Other Names: TBI
Other: Magnetic Affinity Cell Sorting — Device
  Other Names: Magnetic-Activated Cell Sorter (CliniMACS, Miltenyi)
Procedure: Peripheral Blood Stem Cell Transplantation — Patient will undergo a PBSC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; Peripheral Blood Progenitor Cell Transplantation; Transplantation; Peripheral Blood Stem Cell
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Patients who are considered appropriate candidates for allogeneic hematopoietic stem cell transplantation
Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation — Patients who are eligible will receive a T Cell-Depleted Hematopoietic Stem Cell Transplantation

SUMMARY:
RATIONALE: Allogeneic hematopoietic stem cell transplant (HSCT) is a treatment that can cure acute leukemia and myelodysplasia. After giving the patient chemotherapy and total body irradiation to stop the growth of cancer and remove the patient's diseased bone marrow, healthy stem cells from a donor are infused into the patient to replace the patient's bone marrow and make red and white blood cells and platelets. Unfortunately HSCT is often complicated by 'graft versus host disease' (GVHD) in which the transplanted cells from a donor can make an immune response against the body's normal cells and cause tissue damage and severe symptoms. Removing a subset of the donor T cells, called 'naive T cells', before transplant may reduce the frequency and intensity of GVHD.

PURPOSE: This phase II trial will determine whether the removal of the naive T cells from donor cells can decrease the rate and severity of graft-vs-host disease while preserving specific immunity against infections in patients with acute leukemia or advanced myelodysplastic syndromes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the probability of grades II-IV acute graft-vs-host disease (GVHD) in patients with acute leukemia or advanced myelodysplastic syndromes treated with CD45RA+ T-cell-depleted allogeneic peripheral blood stem cell transplantation and compare this to relevant historical experience.
* Estimate the probability of graft failure in these patients.

Secondary

* Evaluate immune reconstitution and pathogen-specific T-cell reconstitution in these patients.
* Estimate the probability of transplant-related mortality by day 100 in these patients.
* Estimate the probability of relapse in these patients.
* Estimate the probability and severity of chronic GVHD in these patients.

OUTLINE: This is a multicenter study.

* Myeloablative conditioning regimen: Patients undergo total body irradiation twice daily for 4 days (Days -10 to -7) Patients also receive thiotepa IV over 4 hours for 2 days (Days -6 and -5) and fludarabine phosphate IV over 30 minutes for 5 days (Days -6 to -2.)
* Transplantation: Patients receive a CD34+ enriched allogeneic peripheral blood stem cell (PBSC) product followed by a CD45RA+ T-cell-depleted allogeneic PBSC product on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients will receive Tacrolimus as per cohort 1. If the rate of grade II-IV acute GVHD in the first 35 patients is significantly reduced (compared to historical controls), subsequent patients are enrolled in cohort 2.

  * Cohort 1: Patients receive tacrolimus IV continuously or orally twice daily beginning on day -1 and continuing until day 50, followed by a standard taper in the absence of grade II-IV acute GVHD.
  * Cohort 2: Patients receive tacrolimus IV continuously or orally twice daily beginning on day -1 and continuing until day 30, followed by a rapid taper in the absence of grade II-IV acute GVHD.

Patients are followed actively for at least 1 year post transplant.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute lymphocytic leukemia (ALL) or acute myeloid leukemia (AML) in first or subsequent remission
  * ALL or AML in relapse or primary refractory ALL or AML with a circulating blast count ≤ 10,000/mm^3
  * Refractory anemia with excess blasts (RAEB) (RAEB-1 or RAEB-2) if the patient has received induction chemotherapy within the past 60 days
* Appropriate candidate for allogeneic hematopoietic stem cell transplantation (HSCT)
* No CNS involvement refractory to intrathecal chemotherapy and/or standard cranial-spinal radiotherapy

PATIENT CHARACTERISTICS:

* Age 14-55
* Creatinine < 1.5 mg/dL
* Cardiac ejection fraction > 45%
* DLCO corrected > 60% of predicted
* Total bilirubin < 2 times upper limit of normal (ULN) (unless attributed to Gilbert syndrome)
* AST and ALT < 2 times ULN
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after transplantation
* HIV negative
* No co-existing disease (other than leukemia or RAEB) that would limit life expectancy to < 3 months
* No uncontrolled infection that, in the opinion of the consulting infectious disease physician, would contraindicate myeloablative HSCT
* No other medical condition that would contraindicate HSCT
* No known hypersensitivity to tacrolimus

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior HSCT
* No concurrent participation in other experimental studies for the prevention of graft-vs-host disease

DONOR CHARACTERISTICS:

* Genotypic or phenotypic HLA-identical related donor
* Able to donate peripheral blood stem cells
* Age > 14 years
* Applicable to male patients only: No female donors who have previously given birth to a male child or have had a pregnancy beyond the first trimester miscarriage or termination of pregnancy or nursing
* No donors who have received blood transfusions
* No CD45 Mutation with aberrant CD45RA isoform expression

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12-17 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bleakley, MD, Principal Investigator — Fred Hutchinson Cancer Center; Warren Shlomchik, MD, Principal Investigator — Yale University School of Medicine/Yale New Haven Hospital
Locations (2):
- United States (2):
  - Yale University School of Medicine/Yale New Haven Hospital, New Haven, Connecticut
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Bleakley M, Sehgal A, Seropian S, Biernacki MA, Krakow EF, Dahlberg A, Persinger H, Hilzinger B, Martin PJ, Carpenter PA, Flowers ME, Voutsinas J, Gooley TA, Loeb K, Wood BL, Heimfeld S, Riddell SR, Shlomchik WD. Naive T-Cell Depletion to Prevent Chronic Graft-Versus-Host Disease. J Clin Oncol. 2022 Apr 10;40(11):1174-1185. doi: 10.1200/JCO.21.01755. Epub 2022 Jan 10. PMID 35007144
- [Derived] Bleakley M, Heimfeld S, Loeb KR, Jones LA, Chaney C, Seropian S, Gooley TA, Sommermeyer F, Riddell SR, Shlomchik WD. Outcomes of acute leukemia patients transplanted with naive T cell-depleted stem cell grafts. J Clin Invest. 2015 Jul 1;125(7):2677-89. doi: 10.1172/JCI81229. Epub 2015 Jun 8. PMID 26053664

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 2 academic medical centers between Dec 2009 and Oct 2014. The first patient was enrolled on December 17, 2009 and the last participant was enrolled in October 2014
Groups:
- Overall Study Participants: CD34+ enriched allogeneic peripheral blood stem cells (PBSC) followed by CD45RA+ T-cell-depleted allogeneic PBSC and tacrolimus for GVHD prophylaxis
Period: D0 to D100 Post-transplant
Arm/Group | Overall Study Participants
Started | 41
Completed | 39
Not Completed | 2
Not completed — Death | 2
Period: D101 to 2 Years Post-transplant
Arm/Group | Overall Study Participants
Started | 39
Completed | 31
Not Completed | 8
Not completed — Death | 8
Period: 2 Years to 5 Years Post-transplant
Arm/Group | Overall Study Participants
Started | 31
Completed | 28
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Participants: CONDITIONING: Patients receive TBI twice per day on days -10 to -7, then thiotepa IV administered over approximately 4 hours on days -6 and -5, and fludarabine IV administered over 30 minutes on days -6 to -2.
  DONOR BONE MARROW TRANSPLANTATION: GCSF-mobilized CD34 enriched PBSC and CD45RA depleted cells infused on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Ptients receive tacrolimus beginning on day -1 by continuous IV infusion, converting to oral formulation when oral feeding is established. If there is no evidence of grade II-IV acute GVHD prior to day 50, tacrolimus is then tapered.
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 37.7 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Graft-vs-host Disease (GVHD): Grade I-IV, Including Those With no Reportable Acute GVHD
Description: Number of participants with aGVHD and severity of aGVHD within the first 360 days post-transplant as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. Acute GVHD is graded by standard criteria, and all suspected cases of acute GVHD will be confirmed histologically by biopsy of an affected organ. The severity of acute GVHD is determined by an assessment of the degree of involvement of the skin, liver, and gastrointestinal tract. Grade I is characterized as mild disease, Grade II as moderate, Grade III as severe (involvement of any organ system), and Grade IV as life-threatening.
Time Frame: Within 360 days of transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 41
Participants
  No acute GVHD | 11
  Grade I acute GVHD | 2
  Grade II acute GVHD | 25
  Grade III acute GVHD | 3
  Grade IV acute GVHD | 0
  Steroid refractory acute GVHD | 0

2. Primary Outcome: Number of Participants Who Did Not Engraft After Receiving a CD45RA+ T Cell Depleted PBSC Transplant
Description: Graft failure is defined as either a failure to reach an ANC of >500/uL for 3 consecutive days by day 28 post-transplant, or an irreversible decrease in ANC <100 after an established donor graft, unless there is a reasonable explanation such as a viral infection or drug effect that may be responsible for a reversible decrease in ANC.
Time Frame: Up to 5 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 41
Participants | 0

3. Secondary Outcome: Transplant-related Mortality by Day 100
Description: Number of participants who died due to transplant-related issues within the first 100 days of transplant
Time Frame: Transplant to day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 41
Participants | 2

4. Secondary Outcome: Number of Participants Who Have Relapsed Within 5 Years of CD45RA+ T Cell Depleted PBSC Transplant
Description: Relapse is defined by the presence of malignant cells in marrow, peripheral blood, or extramedullary sites by histopathology. Testing for recurrent malignancy in the blood and bone marrow performed by monitoring the CBC and bone marrow at Day 28, 58, 80, 360, and as needed for suspected relapse.
Time Frame: Up to 5 years post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 41
Participants | 10

5. Secondary Outcome: Number of Participants With Chronic GVHD
Description: Chronic GVHD measured by meeting NIH criteria and treated with immune suppression
Time Frame: Up to 5 years post transplant
Population: Participants alive and without relapse at D100
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study Participants
Number analyzed (Participants) | 38
Participants
  Chronic GVHD that meets NIH criteria | 3
  No documented chronic GVHD | 35

ADVERSE EVENTS:
Time Frame: AEs and SAEs: Conditioning through Day 100; All-Cause Mortality: Conditioning through 5 year
Description: No Serious Adverse Events reported were related to the investigational cell product, but to the transplant or other indications.
Arm/Group | Overall Study Participants
All-Cause Mortality (participants affected / at risk) | 13/41
Serious Adverse Events (participants affected / at risk) | 39/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study Participants (N=41)
Abdominal pain (Gastrointestinal disorders) | 2 (2) — Grade 3
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) — Grades 2-4
Anorexia (Metabolism and nutrition disorders) | 3 (3) — Grade 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Bladder infection (Infections and infestations) | 2 (2) — Grade 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) — Grade 4
Catheter related infection (Infections and infestations) | 9 (9) — Grade 3
Colitis (Gastrointestinal disorders) | 1 (1) — Grade 3
Dehydration (Metabolism and nutrition disorders) | 3 (3) — Grade 3
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3
Duodenal infection (Infections and infestations) | 1 (1) — Grade 3
Enterocolitis (Gastrointestinal disorders) | 1 (1) — Grade 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 3
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) — Grade 3
Generalized muslce weakness (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Headache (Nervous system disorders) | 1 (1) — Grade 3
Hypotension (Vascular disorders) | 7 (7) — Grades 3-4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) — Grades 3-4
Coagulase-negative staph bacteremia (Infections and infestations) | 8 (8) — Grade 3
Clostridium difficile infection (Infections and infestations) | 3 (3) — Grade 3
CMV reactivation (Infections and infestations) | 20 (20) — Grade 3
E Coli Bacteremia (Infections and infestations) | 2 (2) — Grade 3
Leptotrichia buccalis infection (Infections and infestations) | 1 (1) — Grade 3
MRSA bacteremia (Infections and infestations) | 1 (1) — Grade 3
Candida Glabrata (Infections and infestations) | 1 (1) — Grade 3
Enterococcus faecium (Infections and infestations) | 1 (1) — Grade 3
Strep mitis (Infections and infestations) | 2 (2) — Grade 3
Strep Viridans (Infections and infestations) | 2 (2) — Grade 3
VRE bacteremia (Infections and infestations) | 2 (2) — Grade 3
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 4
Lung infection (Infections and infestations) | 2 (2) — Grade 3
Mucositis, oral (Gastrointestinal disorders) | 36 (37) — Grade 3
Nausea (Gastrointestinal disorders) | 3 (3) — Grade 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — bilateral LE leg pain requiring PCA - Grade 3
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 2 (2) — Grade 3
Pericardial effusion (Cardiac disorders) | 1 (1) — Grade 4
Pericarditis (Cardiac disorders) | 1 (1) — Grade 4
Rectal pain (Gastrointestinal disorders) | 1 (1) — Grade 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 5
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 4
Sepsis (Infections and infestations) | 3 (3) — Grade 4
Sinusitis (Infections and infestations) | 1 (1) — Grade 3
Neutrophil count decreased (Investigations) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study Participants (N=41)
Anemia (Blood and lymphatic system disorders) | 8
Lymphocyte count decreased (Investigations) | 34
Neutrophil count decreased (Investigations) | 16
Platelet count decreased (Investigations) | 13
White blood cell decreased (Investigations) | 15
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 6
CD4 lymphocytes decreased (Investigations) | 33
Diarrhea (Gastrointestinal disorders) | 19
Hypertenstion (Vascular disorders) | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 8 — Grade 3
Anorexia (Metabolism and nutrition disorders) | 5 — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT00914940/Prot_SAP_000.pdf